CLINICAL TRIAL: NCT02634749
Title: OTIS - Optimized Complementary Feeding Study
Acronym: OTIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Semper AB (Unknown); University of California (Other); MRC Human Nutrition Research (Other Government)
Responsible Party: Principal Investigator, Torbjörn Lind, Associate Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Umu_2014-363-31
Record Dates: First submitted 2015-09-30; First posted 2015-12-18 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Infant Development; Body Composition, Beneficial; Dietary Modification
Keywords: Nordic countries; Eating behavior; Human microbiome; Child nutrition; Metabolic profile; Body composition
MeSH Terms: conditions — Glucocorticoid Receptor Deficiency; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nordic diet (Experimental): The participant in the Nordic diet group will experience three interventions: a) a systematic introduction of taste portions, b) Protein reduced complementary foods (milk cereal drinks, porridge and baby milk with reduced protein content), and c) homemade and industry manufactured main meals with a predominance of Nordic ingredients.
  Interventions: Other: Systematic introduction of taste portions; Other: Protein reduced complementary foods; Other: Nordic diet
- Regular diet (No Intervention): The participants will be given the current advice on infant feeding issued by the Swedish National Food Agency. They will also be given regular, commercially available milk cereal drinks, porridge, baby milk and industry manufactured main meals. No advice or recipes on meals will be given apart from the current recommendations.

INTERVENTIONS:
Other: Systematic introduction of taste portions — A systematic introduction of plant foods from the Nordic diet
  Arms: Nordic diet
Other: Protein reduced complementary foods — Specially prepared, protein-reduced, age-adjusted milk cereal drinks, baby cereals and baby milk, and commercially available baby foods in glass jars
  Arms: Nordic diet
Other: Nordic diet — Taste portions, homemade and industry manufactured main meals with a predominance of Nordic ingredients
  Arms: Nordic diet

SUMMARY:
Dietary factors during infancy, e.g. high intakes of protein, fast carbohydrates and saturated fat increase the risk of adult obesity, type 2 diabetes and hypertension. However, current dietary recommendations to infants are based on traditions and experiences whereas research is basically lacking.

Towards the end of the first year of life the infant will normally become increasingly suspicious towards fruits and vegetables. However, these foods are an important part of healthy eating. When and how these food items should be introduced into the diet of young children is unclear.

New Nordic Diet, an initiative from the Nordic Council of Ministers calls for a larger intake of fruits, vegetables, whole grain, fish and game. In adults such diet improves weight and biomarkers of insulin resistance and cardiovascular disease. Since dietary preferences are founded early in life it is logical to introduce such a diet already when the child is starting complementary foods.

In a randomized controlled study from 6 mo of age, we want to explore if a Nordic complementary diet with lower protein intake, more vegetable fats and a systematic introduction of fruits and greens will improve body composition, metabolic biomarkers, the composition of faecal microbiota (associated with obesity), cognitive development and the consumption of foods that can lay the foundation for better long-term diet. If the study has the expected results, these will have a direct impact on the dietary habits of Swedish children during infancy and childhood and thus their long-term health.

DETAILED DESCRIPTION:
Introduction Evidence is accumulating that early feeding affects health and development later in life. The positive effects of breast feeding are well known, but less is known on how different types and timing of complementary foods, i.e. the foods used during the transition from breastfeeding or formula-feeding to family foods affect short and long-term health. During the time of complementary feeding, the demands for energy and nutrients remain high, especially during the second half of the first year of life. We and others have shown a link between protein intake during this time period and later risk for overweight. Earlier studies have implicated very high protein intakes during infancy but the latest dietary recommendations for infants and children suggest lower intakes, which may have contributed to the decreasing prevalence of obesity seen in some countries. Early introduction of carbohydrate-rich complementary foods has also been associated to alterations leading to later obesity and insulin resistance. Finally, we and others have shown that higher intakes of polyunsaturated fatty acids and lower intakes of saturated fatty acids in the diet of infants improve blood lipids and that these influences track into childhood.

The composition of the complementary food is important also from the perspective of food flavour, texture and presentation. Experiences of flavour during foetal and breast feeding period prime the newborn infant to accept the same types of foods as the mother usually takes, including foods with flavours outside the normal preferences of the infant, i.e. sweet, salty and fatty. Also the acceptance of different textures of foods changes during the infancy year. As the oral motor skills of the infant develop, the child is able to handle increasingly lumpy and solid foods. A normally developing infant will have periods of greater acceptance of novel foods both in terms of flavour and texture, usually coinciding with the time when complementary foods are introduced. However, this window of opportunity to introduce new foods begins to close around 10-12 mo. of age, when the child grows increasingly suspicious of unfamiliar tastes, i.e. food neophobia, but also, if solids haven't been introduced at this time, to the texture of common food items. Studies have shown that the types and numbers of different foods that a child accepts can be influenced by the manner and frequency of how they are introduced during this time. Numerous studies have shown that fruits and vegetables are an important part of healthy eating habits in all ages, but that the actual intake of these food items among young children is low. Instead, population-based studies from Sweden have shown that the dietary intake of children is not satisfactory from a public health perspective, with intakes of refined sugars, fatty foods and salt being too high and intakes of fruits and vegetables being too low.

In 2005 the Nordic Council of Ministers launched the New Nordic Food programme. This initiative highlights the health, gastronomic and sustainability aspects of foods produced within the Nordic region. Compared to the regular Swedish diet, the Nordic diet (ND) stresses higher intakes of regionally produced fruits, berries, vegetables, tubers, and legumes, higher intakes of whole-wheat, vegetable fats and oils, fish and egg, and lower intake of sweets, desserts and dairy, meat and poultry products, but at the same time being in line with current dietary recommendations. In adults, studies on ND have shown beneficial effects on weight and metabolic and cardiovascular disease markers of the same magnitude as e.g. the Mediterranean diet.

We aim to improve body composition, metabolic markers and the faecal microbiota composition of young children by using ND as a basis for complementary foods, with its emphasis on regionally produced fruits, berries, vegetables, tubers and legumes, also increasing the intake of fish and vegetable fats and oils, particularly using rapeseed oil but decreasing total protein intake. Effects on faecal microbiota composition have been a proposed pathway linking early dietary intake with later metabolic outcomes.

Relevance The early diet has longstanding effects on human health. Apart from breastfeeding little is known on which infant diets would confer long-term health benefits. ND has several potential advantages in this respect, and studies in adults have shown favourable effects on metabolic and cardiovascular disease markers and mortality similar to those gained through the Mediterranean diet. The present study, using ND as the basis for complementary foods but also reducing the total protein intake, improving fatty acid composition and expanding the introduction of fruits and vegetables into the diet of small children is the first study of its kind and will add vital information in the search to prevent obesity, dyslipidaemia, insulin resistance, type 2 diabetes, hypertension and cardiovascular disease and will have implications for future national and international dietary recommendations to young children. Through early intervention, i.e. already when complementary foods are introduced into the diet of the infant, we believe that we can initiate healthy food preferences from the earliest date thus maximizing the long-term public health benefits of healthy eating. By adopting the concept of ND we will also add gastronomical aspects to the development of optimal complementary foods as well as support regional food production and contribute to a sustainable environment.

Objectives The overall aim of the study is to compare the effects of a ND portfolio intervention on body composition, metabolic markers, blood pressure and faecal microbiota composition to conventional complementary feeding from 6-18 months of age.

More specifically, we will investigate if:

1. A complementary diet lower in protein (total reduction 30%) will affect growth, body composition, i.e. reduce total body fat mass and improve metabolic markers, i.e. decrease plasma (P) levels of insulin, glucose and insulinlike growth factor 1 (IGF1) without detrimental effects on linear growth.
2. A complementary diet based on Nordic foods will affect growth, body composition, i.e. reduce body fat mass and improve metabolic markers and the faecal microbiota composition, i.e. a microbiota composition associated with less obesity and inflammation without detrimental effects on linear growth.
3. Complementary foods with a modified fat intake, i.e. a higher intake of LCPUFA through an increased intake of fish and substituting fats and oils found in regular complementary foods with milk fat and rapeseed oil will improve body composition, metabolic markers, cognitive development and the faecal microbiota composition without detrimental effects on linear growth.
4. A systematic introduction of plant foods from the Nordic diet during weaning will increase the acceptance of new fruits and vegetables into the diet of the young child.

Methods Participants and recruitment Healthy, full-term singletons will be recruited at 4 months of age. When parents consider it appropriate to introduce complementary foods into the diet of their child, but no later than at 6 mo. of age, the child will be randomly allocated to one of two study groups, i.e. the Nordic diet group (intervention, ND) or the Regular diet group (control). The group allocation will be masked for the participants and researchers.

Study products All participants will be provided with study products free of charge. In the ND group these will be specially prepared, protein-reduced, age-adjusted milk cereal drinks (MCDs), baby cereals and baby milk, and commercially available baby foods in glass jars (BIG). The control group will be offered commercially available, age-adjusted MCDs, baby cereals, baby milk and BIG. All products will be manufactured by Semper AB, Sweden.

Introduction of complementary feeding The ND group will be given recipes of fruit and vegetable purees and instructions how to prepare these recipes. The main ingredients will be fruits, berries and vegetables which grow and are available in the Nordic region according to a predefined list. These taste meals will be given to the participating infant when the parents judge it prudent to start offering the infant other foods beside breast milk or formula and the infant is deemed ready by the parent.

The control group will be given the standard, oral and written advice that is given from well-baby clinics to parents when beginning with small taste meals.

Parental support Parents with children in the ND group will be given support to continue following the dietary intervention through social media (Face book). In this forum parents can discuss with the study dietician and among themselves, sharing experiences. Parents will also have instructional videos on the preparation of certain study foods and recipes. Participants will share experiences and other information at their own discretion. No data will be collected through this group, but the group may function as a way to inform the families on the group on upcoming study events and remind participants to send in e.g. questionnaires. Both the intervention and the control group will get monthly telephone calls from the research nurse or the study dietician.

Data collection Main data collection points will be at baseline, i.e. when the child is between 4-6 months of age, and at 9, 12 and 18 months of age. At these time points the participants will come to the Paediatric Research Unit for measurements and sampling.

Procedures The baseline visit and the 9mo. visits will take place at the Paediatric Research Unit at the Department of Clinical Sciences, Paediatrics, Umeå University Hospital (Figure). At ages 7, 8, 10, 11 and 13-17 mo. the research nurse or dietician will have a telephone follow-up with the participants checking adherence, possible study related problems, supply and consumption of study products and the symptoms registrations. At 12 and 18 mo. the participants will again come to the Paediatric Research Unit for samples. Also, the research nurse will do home visits for anthropometric measurements, TBW and the two videotaped tests, i.e. food acceptance test and the free play test.

Informed consent and withdrawal A written Informed Consent from the subject's parents/caregiver is an inclusion criterion without which the subject cannot be included in the study. The participants may withdraw from the study at any time by withdrawing consent, through noncompliance or if the participant experiences adverse events requiring the participant to withdraw on advice of the research physician or by his/her own accord. If possible the reasons for withdrawal will be recorded. Participants that are withdrawn will not be replaced.

D. Statistical analyses and ethical clearance Comparisons of differences in main outcomes between the ND and control groups will be the focus of the statistical analyses. The primary outcomes will be analysed according to the intention-to-treat principle when comparing the two study groups, but per protocol analyses will also be done. Both parametric and nonparametric tests will be used depending on the distribution of data. Possible effect modifiers and confounders will be included in the analyses as needed to explain group differences. Data on dietary intake will be converted to energy and nutrients through nutrient calculation software (Dietist NET, Kost och Näringsdata AB, Bromma, Sweden). The study has ethical clearance from the Regional Ethics committee, Umeå University (Dnr 201436331M).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, singleton infants 4-6 mo. of age
* >37 weeks of gestation at birth
* Birth weight >2500 g
* Available throughout the study period, i.e. the participant will remain in the study area (Umeå municipality) and will not commence child care outside the home during the extent of the study, i.e. until 18 mo. of age.
* Parents or legal guardians are able to give written informed consent to participation in the study.

Exclusion Criteria:

* Children with chronic illnesses that will affect feeding or growth, including food allergies or intolerance to study products
* Intake of any complementary food at recruitment
* Use of supplements or medications that will affect the study outcomes
* Iron deficiency (Hb <105 g/L, S-ferritin <12 µg/L) or any other biochemical abnormality discovered at the baseline examination that needs medical attention after decision by the study physician.
* Repeated non-adherence to key study procedures including anthropometric measurements, allergy, eczema and symptoms registrations

Ages: 4 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Body composition | 12 mo. of age
  Total body water (TBW) as a measure of body composition (3 compartment model) will be determined at 12 months of age. TBW will be assessed using deuterium (2H2O) in collaboration with the MRC Human Nutrition Research Laboratory, Cambridge, UK.
Body composition | 18 mo. of age
  Total body water (TBW) as a measure of body composition (3 compartment model) will be determined at 18 months of age. TBW will be assessed using deuterium (2H2O) in collaboration with the MRC Human Nutrition Research Laboratory, Cambridge, UK.

SECONDARY OUTCOMES:
Dietary intake | 9 mo. of age
  At 9 mo. of age the parents will be asked to register the participating child's intake of foods and drinks during consecutive 5 days.
Dietary intake | 12 mo. of age
  At 12 mo. of age the parents will be asked to register the participating child's intake of foods and drinks during consecutive 5 days. They will also be asked to photograph the child's meal portions just before the meal is served and right after, taking 2 photos each time from perpendicular angles.
Dietary intake | 18 mo. of age
  At 18 mo. of age the parents will be asked to register the participating child's intake of foods and drinks during consecutive 5 days. They will also be asked to photograph the child's meal portions just before the meal is served and right after, taking 2 photos each time from perpendicular angles.
Biomarkers of adherence | 9 mo. of age
  Blood samples will be collected for haemoglobin, iron status, P-urea, vitamins C, A, E, carotenoids, folic acid, cow's milk specific C15 and C17 fatty acids as secondary outcomes and markers of adherence.
Biomarkers of adherence | 12 mo. of age
  Blood samples will be collected for haemoglobin, iron status, P-urea, vitamins C, A, E, carotenoids, folic acid, cow's milk specific C15 and C17 fatty acids as secondary outcomes and markers of adherence.
Biomarkers of adherence | 18 mo. of age
  Blood samples will be collected for haemoglobin, iron status, P-urea, vitamins C, A, E, carotenoids, folic acid, cow's milk specific C15 and C17 fatty acids as secondary outcomes and markers of adherence.
Allergy and atopic manifestations | 9 mo. of age
  At 9 mo. of age the participants will in a questionnaire be asked for symptoms of allergy, asthma, atopic disease and eczema.
Allergy and atopic manifestations | 12 mo. of age
  At 12 mo. of age the participants will in a questionnaire be asked for symptoms of allergy, asthma, atopic disease and eczema.
Allergy and atopic manifestations | 18 mo. of age
  At 18 mo. of age the participants will in a questionnaire be asked for symptoms of allergy, asthma, atopic disease and eczema.
Psychological development (ASQ) | 12 mo. of age
  The Ages and Stages Questionnaire (ASQ) will be administered at 12 mo. of age as a measure of general development.
Psychological development (free play) | 12 mo. of age
  A videotaped single object free play task, as a measurement of cognitive development in relation to the nutritional intervention will be administered at 12 mo. of age.
Psychological development (ASQ) | 18 mo. of age
  The Ages and Stages Questionnaire (ASQ) will be administered at 18 mo. of age as a measure of general development.
Psychological development (free play) | 18 mo. of age
  A videotaped single object free play task, as a measurement of cognitive development in relation to the nutritional intervention will be administered at 18 mo. of age.
Biomarkers of metabolic function | 9 mo. of age
  Blood and urine samples will be collected for a number of biomarkers associated with metabolic function including plasma (P-) insulin, P-glucose, P-IGF-1, P-lipids and lipoproteins, P-fatty acids including LC-PUFAs (DHA, EPA, ARA), hsCRP, oxidative capacity, metabolomics and lipidomics.
Biomarkers of metabolic function | 12 mo. of age
  Blood and urine samples will be collected for a number of biomarkers associated with metabolic function including plasma (P-) insulin, P-glucose, P-IGF-1, P-lipids and lipoproteins, P-fatty acids including LC-PUFAs (DHA, EPA, ARA), hsCRP, oxidative capacity, metabolomics and lipidomics.
Biomarkers of metabolic function | 18 mo. of age
  Blood and urine samples will be collected for a number of biomarkers associated with metabolic function including plasma (P-) insulin, P-glucose, P-IGF-1, P-lipids and lipoproteins, P-fatty acids including LC-PUFAs (DHA, EPA, ARA), hsCRP, oxidative capacity, metabolomics and lipidomics.
Faecal microbiota composition | 12 mo. of age
  Overall faecal microbiota composition using 16S rDNA analysis
Oral microbiota composition | 12 mo. of age
  Overall oral microbiota composition using 16S rDNA analysis
Faecal microbiota composition | 18 mo. of age
  Overall faecal microbiota composition using 16S rDNA analysis
Oral microbiota composition | 18 mo. of age
  Overall oral microbiota composition using 16S rDNA analysis
Blood pressure | 12 mo. of age
  Blood pressure will be measured with the child sitting in the parent's lap using a Carescape Dinamap V100 monitor (GE Healthcare AB, Sweden) and age appropriate blood pressure cuffs. At baseline, the parents' blood pressure will be collected sitting, using the same equipment as described above.
Blood pressure | 18 mo. of age
  Blood pressure will be measured with the child sitting in the parent's lap using a Carescape Dinamap V100 monitor (GE Healthcare AB, Sweden) and age appropriate blood pressure cuffs. At baseline, the parents' blood pressure will be collected sitting, using the same equipment as described above.
Acceptance of test meal | 12 mo. of age
  A video-taped test meal to assess acceptability of new foods will be administered at 12 mo. of age. During the meal the parent will serve a mid-day snack (a fruit-flavoured yoghurt, a fruit-flavoured milk and a cracker with a vegetable spread) to the child.
Acceptance of test meal | 18 mo. of age
  A video-taped test meal to assess acceptability of new foods will be administered at 18 mo. of age. During the meal the parent will serve a mid-day snack (a fruit-flavoured yoghurt, a fruit-flavoured milk and a cracker with a vegetable spread) to the child.
Body mass index | 12 mo. of age
  Body mass index will be calculated from weight and length and assessed at 12 mo. of age
Body mass index | 18 mo. of age
  Body mass index will be calculated from weight and length and assessed at 18 mo. of age

OTHER OUTCOMES:
Prevalence of bitter taste receptor gene hTAS2R28 | Baseline
  Saliva samples at baseline
Temperament | 18 mo. of age
  Child temperament will be assessed with the Swedish versions of the Toddler Behaviour Questionnaire (TBQ) at 18 mo. of age.

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Lind, Ass prof, Principal Investigator — Umeå University
Locations (1):
- Paediatrics, Department of Clinical Sciences, Umeå, Sweden

REFERENCES:
- [Derived] Johansson U, Ohlund I, Lindberg L, Hernell O, Lonnerdal B, Venables M, Lind T. A randomized, controlled trial of a Nordic, protein-reduced complementary diet in infants: effects on body composition, growth, biomarkers, and dietary intake at 12 and 18 months. Am J Clin Nutr. 2023 Jun;117(6):1219-1231. doi: 10.1016/j.ajcnut.2023.03.020. Epub 2023 Mar 27. PMID 36990225
- [Derived] Lind T, Johansson U, Ohlund I, Lindberg L, Lonnerdal B, Tennefors C, Hernell O. Study protocol: optimized complementary feeding study (OTIS): a randomized controlled trial of the impact of a protein-reduced complementary diet based on Nordic foods. BMC Public Health. 2019 Jan 31;19(1):134. doi: 10.1186/s12889-019-6466-1. PMID 30704429